CLINICAL TRIAL: NCT05759936
Title: Effects of 4-week Seaweed Supplementation on Menopause Symptoms and Psychological Wellbeing - a Randomised, Placebo-controlled Trial
Brief Title: 4-week Seaweed Supplementation on Menopause Symptoms and Psychological Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Doctor Seaweed (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Project ID 2434
Record Dates: First submitted 2023-02-10; First posted 2023-03-08 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2023-11

CONDITIONS: Menopausal Syndrome; Menopausal Depression

STUDY DESIGN:
Intervention Model Description: Active vs. placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule consumed for 28 days
  Interventions: Other: Placebo
- 500mg seaweed (Experimental): Seaweed capsule consumed for 28 days
  Interventions: Dietary Supplement: 500mg seaweed

INTERVENTIONS:
Dietary Supplement: 500mg seaweed — 4 week supplementation of 1 capsule per day of seaweed
  Arms: 500mg seaweed
Other: Placebo — 4 week placebo supplement of 1 capsule per day
  Arms: Placebo

SUMMARY:
Menopausal symptoms have a substantial effect on quality of life as well as potentially serving as markers for future health. Previous research has suggested that diet can impact menopausal symptoms. Seaweed is marketed as a treatment to alleviate menopause symptoms, but no research has tested whether it is effective in reducing the symptoms and psychological effects associated with menopause.

The aim of this study is to investigate the effects of consuming a seaweed supplement over a 4-week time period on menopausal symptoms and psychological well-being.

DETAILED DESCRIPTION:
Menopause and peri-menopause are associated with a number of symptoms and psychological well-being. Previous literature has found a relationship between diet and menopause management. For example, following the Mediterranean diet consuming a variety of vegetables, fruits, legumes and whole grains has found to improve menopausal symptoms particularly vasomotor symptoms. Few studies have explored the effects of dietary supplements on psychological well-being in menopause. The aim of the study is to explore the impact of an iodine-rich seaweed food supplement on menopause symptoms and mental well-being in those experiencing menopause. Online assessments of symptoms will take place pre-intervention and post-intervention and will be compared to the effects of a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Self-assess as healthy
* Experienced menopausal or peri-menopausal symptoms in the past 6 months

Exclusion Criteria:

* Are currently taking HRT, anti-depressants, or anti-anxiety medication
* Are lactating or pregnant (or seeking to become pregnant)
* Have a thyroid disorder
* Are currently taking iodine supplements
* Have any relevant food intolerances

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
The Menopause-Specific Quality of Life Questionnaire (Hildtich, 1996) | At 28 days post-dose, adjusted for baseline
  The menopause-specific quality of life questionnaire assesses the effect of menopausal symptoms on quality of life in four domains: vasomotor, psychosocial, physical, and sexual; as well as providing a total score. The questionnaire has 29 items, each item is a symptom of menopause, the participants rate each symptom between 0 (not at all bothered) to 6 (bothered all the time.) The physical symptoms include items such as 'hot flushes' and 'sweating'; psychological symptoms include 'accomplishing less than I used to' and 'poor memory'; physical symptoms include 'difficulty sleeping' and 'weight gain'; sexual symptoms include 'vaginal dryness' and 'avoiding intimacy'. A conversion score is created for each of the 4 domains: vasomotor; psychosocial; physical; sexual; as well as a total score. Each score ranges from 1 -8, with higher scores indicating greater problems.
Centre for Epidemiologic Studies Depression Scale (Radlof, 1997) | At 28 days post-dose, adjusted for baseline
  This is an established questionnaire used to measure symptoms associated with depression. The questionnaire has 20 items, including 'my sleep is restless', 'I felt depressed' and 'I felt lonely'. The participants rate the symptom on a scale between <1 day and 5 to 7 days, the 4 scale points are: Rarely or none of the time (less than 1 day); Some or a little of the time (1-2 days); Occasionally or a moderate amount of time (3-4 days); Most or all of the time (5-7 days). The possible range of scores is between 0 to 60, higher scores indicate more presence of symptomatology. The scoring of positive items is reversed.
The State-Trait Anxiety Inventory (Spielberger, 1983) | At 28 days post-dose, adjusted for baseline
  The state-trait anxiety inventory will be used to measure anxiety levels, specifically trait anxiety. It consists of 20 items and the scale ranges from 1 to 4: 1 = almost never, 2 = sometimes, 3 = often and 4 = almost always. The nine positive items will be reversed for scoring, items 21, 23, 26, 27, 30, 33, 34, 36 and 39. The possible range of scores is 20 to 80, higher scores indicate higher levels of trait anxiety within the participant. Examples of items within the questionnaire include: 'I feel like a failure' and 'I feel secure'.
The Perceived Stress Scale (Cohen et al., 1983) | At 28 days post-dose, adjusted for baseline
  This established questionnaire will be used to measure the perception of stress. Each of the ten items are rated on a scale between 0 (never) to 4 (very often.) The five scale points are 0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often. The four positive items will be reversed for scoring, items 4, 5, 7 and 8. The questionnaire item examples include 'In the last month, how often have you been upset because of something that happened unexpectedly?' and 'In the last month, how often have you felt that you were unable to control the important things in your life?'. The possible range of scores is between 0 to 40, higher scores indicate high participant perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Haskell-Ramsay, Principal Investigator — Northumbria University
Locations (1):
- Online, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An anonymised dataset will be shared via an open data repository (Open Science Framework). Any information which may identify individual participants will be removed from the dataset before it is shared. Data will be shared in accordance with FAIR (findable, accessible, interoperable, reusable) principles. Participants will consent to the data being shared in this way
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 3 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Fully accessible